CLINICAL TRIAL: NCT03134222
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Filgotinib and GS-9876 in Female Subjects With Moderately-to-Severely Active Cutaneous Lupus Erythematosus (CLE)
Brief Title: Study to Evaluate Safety and Efficacy of Filgotinib and Lanraplenib in Females With Moderately-to-Severely Active Cutaneous Lupus Erythematosus (CLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-436-4092
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lanraplenib 30 mg (Experimental): Lanraplenib + filgotinib placebo for 48 weeks
  Interventions: Drug: Lanraplenib; Drug: Filgotinib placebo
- Filgotinib 200 mg (Experimental): Filgotinib + lanraplenib placebo for 48 weeks
  Interventions: Drug: Filgotinib; Drug: Lanraplenib placebo
- Placebo (Placebo Comparator): Filgotinib placebo + lanraplenib placebo for 12 weeks
  Interventions: Drug: Lanraplenib placebo; Drug: Filgotinib placebo
- Placebo to Lanraplenib 30 mg (Experimental): After Week 12 Visit, participants on placebo will be rerandomized 1:1 and receive lanraplenib + filgotinib placebo in a blinded fashion through Week 48.
  Interventions: Drug: Lanraplenib; Drug: Filgotinib placebo
- Placebo to Filgotinib 200 mg (Experimental): After Week 12 Visit, participants on placebo will be rerandomized 1:1 and receive filgotinib + lanraplenib placebo in a blinded fashion through Week 48.
  Interventions: Drug: Filgotinib; Drug: Lanraplenib placebo

INTERVENTIONS:
Drug: Lanraplenib — 30 mg tablets administered orally once daily with or without food
  Other Names: GS-9876
  Arms: Lanraplenib 30 mg; Placebo to Lanraplenib 30 mg
Drug: Filgotinib — 200 mg tablets administered orally once daily with or without food
  Other Names: GS-6034
  Arms: Filgotinib 200 mg; Placebo to Filgotinib 200 mg
Drug: Lanraplenib placebo — Tablets administered orally once daily with or without food
  Arms: Filgotinib 200 mg; Placebo; Placebo to Filgotinib 200 mg
Drug: Filgotinib placebo — Tablets administered orally once daily with or without food
  Arms: Lanraplenib 30 mg; Placebo; Placebo to Lanraplenib 30 mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy of filgotinib and lanraplenib (formerly GS-9876) in females with moderately-to-severely active cutaneous lupus erythematosus (CLE).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of CLE, either chronic (e.g., discoid) or subacute CLE per investigator evaluation, with the following:

  * Moderately-to-severely active CLE (Cutaneous lupus erythematosus disease area and severity index [CLASI] activity score ≥ 10) at screening and Day 1
  * Prior intolerance or inadequate response to at least one of the listed medications for the treatment of CLE
* Stable dose (defined as no change in prescription for at least 28 days prior to Day 1) of antimalarials and/or topical or oral corticosteroids is permitted during the study. Individuals who are not planning to continue these medications during the study must have discontinued them at least 28 days prior to Day 1

Key Exclusion Criteria:

* Use of prohibited concomitant medications per study protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (13):
  - Wallace Rheumatic Studies Center, Beverly Hills, California
  - St. Jude Hospital Yorba Linda DBA Dr. Joseph Heritage Healthcare, Fullerton, California
  - Dermatology Research Associates, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - Medderm Associates, San Diego, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Omega Research Consultants LLC, DeBary, Florida
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
- Canada (3):
  - Dermatology Ottawa Research Centre, Ottawa
  - University Health Network (UHN) - Toronto Western Hospital, Toronto
  - K.Papp Clinical Research, Waterloo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Werth VP, Fleischmann R, Robern M, Touma Z, Tiamiyu I, Gurtovaya O, Pechonkina A, Mozaffarian A, Downie B, Matzkies F, Wallace D. Filgotinib or lanraplenib in moderate to severe cutaneous lupus erythematosus: a phase 2, randomized, double-blind, placebo-controlled study. Rheumatology (Oxford). 2022 May 30;61(6):2413-2423. doi: 10.1093/rheumatology/keab685. PMID 34498056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Canada. The first participant was screened on 24 May 2017. The last study visit occurred on 18 December 2019.
Pre-assignment Details: 72 participants were screened.
Groups:
- Lanraplenib 30 mg: Lanraplenib 30 mg + filgotinib placebo tablets orally once daily for 48 weeks
- Filgotinib 200 mg: Filgotinib 200 mg + lanraplenib placebo tablets orally once daily for 48 weeks
- Placebo: Participants received filgotinib placebo + lanraplenib placebo tablets orally once daily for 12 weeks.
- Placebo to Lanraplenib 30 mg: After Week 12 Visit, participants on placebo were rerandomized 1:1 and received lanraplenib 30 mg + filgotinib placebo once daily in a blinded fashion through Week 48.
- Placebo to Filgotinib 200 mg: After Week 12 Visit, participants on placebo were rerandomized 1:1 and received filgotinib 200 mg + lanraplenib placebo once daily in a blinded fashion through Week 48.
Period: Treatment Period (Up to Week 12)
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo | Placebo to Lanraplenib 30 mg | Placebo to Filgotinib 200 mg
Started | 19 | 18 | 10 | 0 | 0
Completed | 14 | 14 | 8 | 0 | 0
Not Completed | 5 | 4 | 2 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 1 | 1 | 0 | 0
Period: Treatment Period (Week 12 to 48)
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo | Placebo to Lanraplenib 30 mg | Placebo to Filgotinib 200 mg
Started | 14 | 14 | 0 (Participants were rerandomized 1:1 to either Placebo to Lanraplenib or Placebo to Filgotinib arm.) | 4 (Participants were rerandomized from the Placebo arm.) | 4 (Participants were rerandomized from the Placebo arm.)
Completed | 12 | 11 | 0 | 3 | 3
Not Completed | 2 | 3 | 0 | 1 | 1
Not completed — Withdrew Consent | 0 | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants received filgotinib placebo + lanraplenib placebo tablets orally once daily for 12 weeks. After Week 12 Visit, participants were rerandomized 1:1 and received filgotinib 200 mg + lanraplenib placebo or lanraplenib 30 mg + filgotinib placebo once daily in a blinded fashion through Week 48.
- Total: Total of all reporting groups
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo | Total
Number analyzed (Participants) | 19 | 17 | 9 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.0) | 43 (11.5) | 46 (7.3) | 47 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 9 | 45
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Black | 6 | 8 | 1 | 15
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  White | 12 | 7 | 6 | 25
  Other | 0 | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 9
  Not Hispanic or Latino | 16 | 13 | 7 | 36
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 1 | 3 | 8
  United States | 15 | 16 | 6 | 37
Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score [Mean (Standard Deviation); unit: score on a scale] — CLASI Activity score ranges from 0-70, higher scores indicate more severe skin disease. For additional details on this index, please see Outcome Measure#1.
  Measure Analysis Population Description: Participants in the Full Analysis Set (who were randomized and received at least one dose of study drug (filgotinib, lanraplenib or placebo) were analyzed.
  score on a scale | 17.1 (6.11) | 19.7 (14.35) | 14.8 (4.79) | 17.6 (9.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score From Baseline to Week 12
Description: CLASI Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and nonscarring alopecia. Evaluation of erythema and scale/hyperkeratosis is based on a table: rows represent anatomical areas and columns represent major clinical symptoms. The extent of involvement for each of the skin symptoms is documented for each anatomic area. The total score ranges from 0-70, with higher scores indicating more severe skin disease.
Time Frame: Baseline; Week 12
Population: Treatment policy-estimand is the primary estimand for the primary endpoint analysis which involved participants in the Full Analysis Set (who were randomized and received at least one dose of study drug [filgotinib, lanraplenib or placebo]) with available data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo
Number analyzed (Participants) | 16 | 16 | 8
score on a scale | -4.5 (1.91) | -8.7 (1.85) | -5.5 (2.56)
Statistical Analysis 1: Comparison: Lanraplenib 30 mg vs Placebo; Test type: Superiority; p = 0.7500, Mixed-effect repeated measures model
Statistical Analysis 2: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; p = 0.3047, Mixed-effect repeated measures model

2. Secondary Outcome: Percentage of Participants at Week 12 With Decrease of ≥ 5 Points in CLASI Activity Score From Baseline
Description: as for outcome 1
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set were analyzed. Missing data are imputed as No Response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo
Number analyzed (Participants) | 19 | 17 | 9
Percentage of participants | 47.4 [24.4 to 71.1] | 64.7 [38.3 to 85.8] | 44.4 [13.7 to 78.8]
Statistical Analysis 1: Comparison: Lanraplenib 30 mg vs Placebo; Test type: Superiority; p = 0.8869, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; p = 0.3293, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants at Week 12 With No Worsening in CLASI Activity Score From Baseline
Description: CLASI Activity is scored based on erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and nonscarring alopecia. Evaluation of erythema and scale/hyperkeratosis is based on a table: rows represent anatomical areas and columns represent major clinical symptoms. The extent of involvement for each of the skin symptoms is documented for each anatomic area. The total score ranges from 0-70, with higher scores indicating more severe skin disease. Worsening was defined as ≥ 3 point increase in CLASI activity score.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set were analyzed. Missing data are imputed as No Response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo
Number analyzed (Participants) | 19 | 17 | 9
Percentage of participants | 84.2 [60.4 to 96.6] | 94.1 [71.3 to 99.9] | 88.9 [51.8 to 99.7]
Statistical Analysis 1: Comparison: Lanraplenib 30 mg vs Placebo; Test type: Superiority; p = 0.7456, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; p = 0.6407, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants at Week 24 With Decrease of ≥ 5 Points in CLASI Activity Score From Baseline
Description: as for outcome 1
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set who were randomized to Filgotinib 200 mg or Lanraplenib 200 mg.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 14 | 12
Percentage of participants | 50.0 [23.0 to 77.0] | 83.3 [51.6 to 97.9]
Statistical Analysis 1: Comparison: Lanraplenib 30 mg; Test type: Other; p < 0.0001, One sample exact binomial test
Statistical Analysis 2: Comparison: Filgotinib 200 mg; Test type: Other; p < 0.0001, One sample exact binomial test

5. Secondary Outcome: Percentage of Participants at Week 24 With No Worsening in CLASI Activity Score From Baseline
Description: as for outcome 3
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set who were randomized to Filgotinib 200 mg or Lanraplenib 200 mg.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 14 | 12
Percentage of participants | 85.7 [57.2 to 98.2] | 100.0 [73.5 to 100.0]
Statistical Analysis 1: Comparison: Lanraplenib 30 mg; Test type: Other; p < 0.0001, One sample exact binomial test
Statistical Analysis 2: Comparison: Filgotinib 200 mg; Test type: Other; p < 0.0001, One sample exact binomial test

ADVERSE EVENTS:
Time Frame: First dose date up to Week 48 plus 30 days
Description: The Safety Analysis Set included participants who received at least one dose of study drug.
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Placebo | Placebo to Lanraplenib 30 mg | Placebo to Filgotinib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17 | 0/9 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/17 | 0/9 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 17/19 | 11/17 | 6/9 | 3/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanraplenib 30 mg (N=19) | Filgotinib 200 mg (N=17) | Placebo (N=9) | Placebo to Lanraplenib 30 mg (N=4) | Placebo to Filgotinib 200 mg (N=4)
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanraplenib 30 mg (N=19) | Filgotinib 200 mg (N=17) | Placebo (N=9) | Placebo to Lanraplenib 30 mg (N=4) | Placebo to Filgotinib 200 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Acne pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03134222/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03134222/SAP_001.pdf